CLINICAL TRIAL: NCT01215773
Title: Pharmacokinetics, Safety and Tolerability of BI 671800 HEA Given 200 mg b.i.d. or 400 mg b.i.d. Over 7 Days. A Randomised, Double Blind, Placebo Controlled Within Dose Groups Phase I Study in Healthy Male and Female Volunteers.
Brief Title: Pharmacokinetics, Safety and Tolerability of BI 671800 HEA Given Over 7 Days. A Randomised, Double Blind, Placebo Controlled Within Dose Groups Phase I Study in Healthy Male and Female Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1268.59; 2009-016369-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-09-29; First posted 2010-10-07 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 671800

ARMS (3):
- BI 671800 HEA medium dose (Experimental): Tablet, oral administration with 240 mL of water for each treatment
  Interventions: Drug: BI 671800
- BI 671800 HEA high dose (Experimental): 2 Tablets, oral administration with 240 mL of water for each treatment
  Interventions: Drug: BI 671800
- Placebo (Placebo Comparator): Matching to HEA 200 mg tablets, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching to HEA 200 mg tablet, oral administration
  Arms: Placebo
Drug: BI 671800 — High dose oral administration
  Arms: BI 671800 HEA high dose
Drug: BI 671800 — Medium dose oral administration
  Arms: BI 671800 HEA medium dose

SUMMARY:
The main objectives of the multiple dose study are to investigate the safety, tolerability pharmacokinetics of BI 671800 HEA in healthy male and female volunteers following multiple oral administration of BI 671800

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age 21 to 50 years (incl.)
3. Body Mass Index (BMI) 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
8. Intake of drugs with a long half life (>24 h) within one month or less than 10 half-lives of the respective drug prior to first study drug administration
9. Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
10. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes daily)
11. Alcohol abuse (average consumption of more than 20 g/day in females and 30 g/day in males) or positive alcohol test
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to day 1 of visit 2)
14. Any laboratory value outside the reference range that is of clinical relevance, especially repeated Alanine transaminase (ALT), Aspartate transaminase (AST), Gamma-glutamyl-transferase (GGT), Alkaline phosphatase (ALP) or total bilirubin above upper limit of normal (ULN) at screening and not resolved before dosing.
15. Inability to comply with dietary regimen of trial site
16. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval within 10 days prior to administration or during the trial, and CYP2C8 substrates such as amiodarone, amodiaquine, paclitaxel, rosiglitazone, pioglitazone and repaglinide or CYP2C9 such as warfarin, tolbutamide, phenytoin, losartan, acenocoumarol within 1 month or six half lives (whichever is greater).
17. Repeated demonstration of a QTc interval >450 ms, PR interval >230 ms or a QRS interval >120 ms; history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)

    For female subjects of childbearing potential only:
18. Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 2 months after study completion
19. No adequate contraception during the study including three months before first dosing until 2 month after study completion, e.g. not any of the following: implants, injectables, combined hormonal contraceptives, intrauterine device, or surgical sterilisation (including hysterectomy). In addition to this, also a barrier method (e.g. condom) will be required, if the female is not surgically sterilised.
20. Lactation

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Vital signs (pulse rate (PR)) | 12 weeks
Clinical laboratory test (clinical chemistry) | 12 weeks
Clinical laboratory test (urinalysis) | 12 weeks
Physical examination | 12 weeks
Vital signs (blood pressure (BP)) | 12 weeks
12-lead ECG (electrocardiogram) | 12 weeks
Clinical laboratory test (haematology) | 12 weeks
Adverse events | 12 weeks
Assessment of tolerability by investigator | 12 weeks

SECONDARY OUTCOMES:
Cmax (maximum plasma concentration of BI 671800 or BI 600957) | up to day 12 post treatment
tmax (time from dosing until maximum concentration of BI 671800 or BI 600957 is measured) | up to day 12 post treatment
AUC0-infinity (area under the plasma concentration-time curve of BI 671800 or BI 600957 from time of dosing extrapolated to infinity) | up to day 12 post treatment
AUCτ,1 (area under the plasma concentration-time curve of BI 671800 or BI 600957 for the complete dosing interval τ) | up to day 12 post treatment
AUC0-tz (area under the plasma concentration-time curve of BI 671800 or BI 600957 from time of dosing to time tz of last quantifiable concentration) | up to day 12 post treatment
Cmax,ss (maximum plasma concentration of BI 671800 or BI 600957 at steady state) | up to day 12 post treatment
tmax,ss (time from dosing until maximum concentration of BI 671800 or BI 600957 at steady state is measured) | up to day 12 post treatment
Cavg,ss (average measured plasma concentration of BI 671800 or BI 600957 at steady state) | up to day 12 post treatment
AUCτ,ss (area under the plasma concentration-time curve of BI 671800 or BI 600957 at steady state for the complete dosing interval τ) | up to day 12 post treatment
λz,ss (terminal rate constant of BI 671800 or BI 600957 in plasma at steady state) | up to day 12 post treatment
t1/2,ss (terminal half-life of BI 671800 or BI 600957 in plasma at steady state) | up to day 12 post treatment
MRTpo,ss (mean residence time of BI 671800 in the body at steady state after oral administration) | up to day 12 post treatment
CL/F,ss (apparent clearance of BI 671800 at steady state following oral administration) | up to day 12 post treatment
Vz/F,ss (apparent volume of distribution of BI 671800 during the terminal phase at steady state following oral administration) | up to day 12 post treatment
RAUCτ,ss,M/P (ratio of AUCτ,ss of the BI 600957 to AUCτ,ss of BI 671800) | up to day 12 post treatment
RCmax,ss,M/P (ratio of Cmax,ss of the BI 600957 to Cmax,ss of BI 671800) | up to day 12 post treatment
accumulation ratios RA,Cmax | up to day 12 post treatment
accumulation ratios RA,AUC | up to day 12 post treatment
peak-trough fluctuation (PTF) of BI 671800 | up to day 12 post treatment
peak-trough fluctuation (PTF) of BI 600957 | up to day 12 post treatment
linearity index (LI) of BI 671800 in plasma | up to day 12 post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1268.59.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany